CLINICAL TRIAL: NCT03632382
Title: Non-invasive Device for the Screening and Diagnosis of Sleep Apnea Syndrome
Acronym: Episas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: SATT Linksium GRENOBLE (Unknown); ARTEHIS (Unknown); ARCTIC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC17.359
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea diagnosis; 3D acquisition
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSA diagnosis with 3D acquisition (Other): OSA diagnosis with 3D acquisition
  Interventions: Diagnostic Test: 3D acquisition of maxillofacial characteristics

INTERVENTIONS:
Diagnostic Test: 3D acquisition of maxillofacial characteristics — A 3D acquisition of maxillofacial characteristics will be performed for each patient in order to validate a predictive model comparable to data obtained by polysomnography

SUMMARY:
This prospective study aims to establish and evaluate a predictive model to diagnose OSA with maxillofacial characteristics 3D acquisition.

DETAILED DESCRIPTION:
Polysomnography is the gold-standard for obstructive sleep apnea (OSA) diagnosis. However, OSA is still undiagnosed. Maxillofacial profile can influence OSA severity. Morphological characteristics can be identified but are not enough measurable and analysable by physicians. 3D acquisition of maxillofacial characteristics with a user-friendly tool, quick and low-priced could be used to obtain a predictive model as an OSA risk indicator. Thus, the aim of this study is to establish and evaluate a predictive model to diagnose OSA with maxillofacial characteristics 3D acquisition.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m²
* caucasian men
* patients from the sleep laboratory (CHU Grenoble Alpes) admitted for a polysomnography
* Patient who has given free and informed consent in writing

Exclusion Criteria:

* history of maxillofacial surgery
* dental malocclusion
* patient involved in another clinical research study
* patient not affiliated with social security
* patient deprived of liberty or hospitalized without consent

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Establish and evaluate a predictive model for OSA diagnosis by 3D acquisition of characteristics maxillofacial | 1 measure at inclusion
  apnea hypopnea index will be measured by polysomnography for each patient and compared to a predictive model establish from body mass index and 3D acquisition (cricomental distance...)

SECONDARY OUTCOMES:
Sensitivity study from different stages of OSA severity | 1 measure at inclusion
  OSA severity stages will be apnea hypopnea index <5, <10, <15
Compare diagnosis performances of predictive model and Berlin or NoSAS questionnaires | 1 measure at inclusion
  Correlation between the Berlin or NoSAS score and the predictive model results
Evaluate performances of the combination (Berlin questionnaire + predictive model) to estimate the OSA risk | 1 measure at inclusion
  Calculate the sensitivity, specificity, predictive positive value and predictive negative value of the combination

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monna F, Ben Messaoud R, Navarro N, Baillieul S, Sanchez L, Loiodice C, Tamisier R, Joyeux-Faure M, Pepin JL. Machine learning and geometric morphometrics to predict obstructive sleep apnea from 3D craniofacial scans. Sleep Med. 2022 Jul;95:76-83. doi: 10.1016/j.sleep.2022.04.019. Epub 2022 Apr 29. PMID 35567881